CLINICAL TRIAL: NCT03359187
Title: Prevention of Radiation-induced Mucositis in Patients With Head and Neck Cancer Treated With Radiotherapy : A Double-blind Randomized Controlled Trial
Brief Title: Prevention of Mucositis in Patients With Head and Neck Cancer Treated With Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulabhorn Hospital (Other)
Responsible Party: Principal Investigator, Sirikorn Rojthamarat, Principle Investigator, Chulabhorn Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 004/2559
Record Dates: First submitted 2016-09-26; First posted 2017-12-02 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Radiation- Induced Mucositis; Adverse Effect of Radiation Therapy; Head and Neck Cancer
Keywords: Radiation- induced mucositis; Head and Neck Cancer; Radiation therapy side effect
MeSH Terms: conditions — Radiation Injuries; Head and Neck Neoplasms | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Experimental design in 3 groups
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Normal saline with salt/Soda (Active Comparator): Normal saline with salt/soda rinse 4 times a day/everyday and for each time 15 ml.
  Interventions: Other: Normal saline with salt/Soda
- Clinacanthus nutans (Experimental): Clinacanthus nutans in form of mouth wash rinse 4 times a day/everyday and for each time 15 ml.
  Interventions: Other: Clinacanthus nutans
- Boesenbergia rotunda (Experimental): Boesenbergia rotunda in form of mouth wash 4 times a day/everyday and for each time 15 ml.
  Interventions: Other: Boesenbergia rotunda

INTERVENTIONS:
Other: Normal saline with salt/Soda — Head and Neck cancer Patients have to rinse 4 times a day/everyday for 15 ml. each time during and after completed the radiation treatment
  Arms: Normal saline with salt/Soda
Other: Clinacanthus nutans — Head and Neck cancer Patients have to rinse 4 times a day/everyday for 15 ml. each time during and after completed the radiation treatment
  Arms: Clinacanthus nutans
Other: Boesenbergia rotunda — Head and Neck cancer Patients have to rinse 4 times a day/everyday for 15 ml. each time during and after completed the radiation treatment
  Arms: Boesenbergia rotunda

SUMMARY:
Prevention of radiation-induced mucositis in patients with head and neck cancer treated with radiotherapy : A Double-blind Randomized Controlled Trial

DETAILED DESCRIPTION:
To compare the effect of each herb extracts in form of mouth wash to protect or delay the onset of the radiation-induced mucositis from the adverse effects of radiation therapy in patients with head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15 years old or older,
* Diagnosed with Head and Neck cancer
* On treatment of external Radiation therapy

Exclusion Criteria:

* Pregnant
* Previously underwent external Radiation therapy
* Illiterate

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change of mucositis grading | Change from baseline mucositis grading 1,2, 3, 4, 5 , 6 , 7, 8, 9 week and at 1 month after completed Radiation therapy
  RTOG (Radiation Therapy Oncology Group) Grade0: none Grade 1 : oral soreness, erythema Grade 2 : oral erythema, ulcer, solid diet tolerated Grade 3 : oral ulcers, liquid diet only Grade 4 : oral alimentation impossible

SECONDARY OUTCOMES:
Patient satisfaction with the mouth wash | The last fraction of radiation therapy, through study completion, an average of 1 year
  Scoring 1-4 not satisfied slightly satisfied moderately satisfied very satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Chulabhorn Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Kongwattanakul S, Petchann N, Petroch P, Thanthong S, Tungfung S, Chamchod S, Pitiporn S, Nantajit D. Prophylactic management of radiation-induced mucositis using herbal mouthwash in patients with head and neck cancer: an assessor-blinded randomized controlled trial. J Complement Integr Med. 2022 Feb 28;19(3):771-780. doi: 10.1515/jcim-2021-0457. eCollection 2022 Sep 1. PMID 35218685